CLINICAL TRIAL: NCT04565457
Title: A Pilot Study Evaluating the Effect of 2D Antiscatter Grids on CBCT Image Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-1684.cc; R01CA245270 (NIH)
Record Dates: First submitted 2020-09-18; First posted 2020-09-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Head and Neck Cancers; Upper Abdomen Cancers
MeSH Terms: conditions — Prostatic Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants Scanned (Experimental): All participants will be scanned with a CBCT system equipped with 2D antiscatter grid technology, referred to as research CBCT. Each participant will also be scanned with a standard clinical CBCT as part of their standard clinical care, which will serve as the baseline, or control.
  Interventions: Device: Research CBCT

INTERVENTIONS:
Device: Research CBCT — Each study participant will receive one additional CBCT scan, with 2D antiscatter grid in place. This is the only intervention in the study, referred as research CBCT scan, and it will be performed on one of the days during the participant's radiation treatment course. This additional research CBCT scan will be used strictly for the objectives of this study. It will not be used as part of the standard clinical care, such as imaging guidance of participant's radiation treatment or diagnostic purposes. To deliver participant's radiation treatment under CBCT guidance, a standard clinical CBCT scan will be acquired, as in standard clinical care protocols.

SUMMARY:
This is Pilot study that investigates the CBCT(Cone beam computed tomography) image quality improvement provided by the 2D antiscatter grid technology. The primary objective is to assess the improvement in tissue visualization in an observer study, which will be conducted in a blinded fashion.

DETAILED DESCRIPTION:
This is a single arm study, where all participants will be scanned with a CBCT system equipped with 2D antiscatter grid technology, referred to as research CBCT. Each participant will also be scanned with a standard clinical CBCT as part of their standard clinical care, which will serve as the baseline, or control. Thus, the image quality improvement in research CBCT will assessed with respect to standard clinical CBCT.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be a male or female aged 18-100.
4. Participants who will be treated or are currently being treated with CBCT-guided photon therapy for prostate or prostate-bed, abdomen head and neck, or pelvic cancers, or with image-guided proton therapy for prostate or prostate bed cancer.

Exclusion Criteria:

1. Metallic implants in the CBCT scan volume, such as hip prostheses or spine stabilization hardware. Patients with pacemakers, defibrillators, or other implanted electronic devices. Dental implants, fillings, or fiducial markers may be acceptable, and the decision for inclusion/exclusion will be on a case-by-case basis, by reviewing prior CT images of the study candidate. Patient's prior CT images will be reviewed by the PI or the site PI.
2. Patients who do not have the ability to lie still for the duration of his/her CBCT imaging and treatment should be excluded. If image artifacts in prior scans are deemed excessive, the patient will be excluded from the study.
3. Known pregnancy. (Per SOC, a pregnancy test will be performed prior to CBCT scan on Day 1. At this time, women of child-bearing potential (WOCBP) will receive a pregnancy test to re-confirm eligibility).

   * Women of child-bearing potential are described as:

     1. Age 55 or younger who have not had a negative pregnancy test within 3 days. This excludes patients who have had tubal ligation or are already post-menopausal.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Change in tissue visualization in CBCT images | 4 years
  IImprovement in image quality and quantitative accuracy as measured by established image quality metrics, such as Hounsfield Unit accuracy, artifact amplitude and contrast-to-noise ratio.

SECONDARY OUTCOMES:
Comparison of tissue delineation in CBCT images by auto-segmentation software. | 4 years
  Similarity of anatomical structures delineated by autosegmentation software and expert observers, , as measured by structure similarity metrics, such as DICE coefficient or Hausdorff distance.

OTHER OUTCOMES:
Concordance Correlation Coefficients | 4 years
  Correlation of radiomics features in CBCT images and gold standard MDCT images, as measured by correlation coefficients, such as Pearson Correlation Coefficient or Concordance Correlation Coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Cem Altunbas, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - University of Florida Health Proton Therapy Institute, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No